CLINICAL TRIAL: NCT06208501
Title: The Predictive Role of Proteomics in Blood Pressure Response of Hypertensive Patients Undergoing Renal Denervation.
Acronym: PREDICT-RDN
Status: Recruiting | Type: Observational
Sponsor: Hippocration General Hospital (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Biomedical Research Foundation, Academy of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Professor, Hippocration General Hospital
Other Study IDs: PREDICT-RDN
Record Dates: First submitted 2023-12-03; First posted 2024-01-17 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Hypertension; Renal Denervation; Proteomics
Keywords: Hypertension; Sympathetic nervous system hyperactivity; Renal denervation; Renal nerves ablation; Proteome; Urine proteomics; Proteomic analysis
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertensive patients undergoing renal denervation
  Interventions: Diagnostic Test: Urine sample for proteomic analysis; Diagnostic Test: ABPM; Diagnostic Test: OBPM

INTERVENTIONS:
Diagnostic Test: Urine sample for proteomic analysis — Urine sample for proteomic analysis in screen visit (before renal denervation procedure).
Diagnostic Test: ABPM — ABPM in screen visit and 3 months after renal denervation procedure.
Diagnostic Test: OBPM — OBPM in screen visit and 3 months after renal denervation procedure.

SUMMARY:
Renal sympathetic nervous activity plays a crucial role in the development and maintenance of hypertension (HTN). Renal denervation (RDN) is a minimally invasive catheter-based treatment using mainly radiofrequency or ultrasound energy to selectively disrupt the sympathetic renal nerves. RDN has experienced rises and falls during its development as a treatment option for HTN in humans. Latest well-designed sham-controlled randomised trials with improved methodology confirmed significant blood pressure (BP) reduction in both office and 24-hour ambulatory BP. Although the safety of RDN procedures seems favourable thus, the rate of BP response to the procedure is variable, with response rates reported in the range between 60% and 70%. It is of great importance to identify biomarkers able to reliably predict subjects who would benefit from this treatment, in order to achieve better therapeutic results.

Proteomics is the study of the full complement of proteins produced or modified by a biological system (cell, tissue, organ, biological fluid, or organism). Proteomic analysis is used in different research settings to understand pathogenicity mechanisms and emerge biomarkers with predictive role in diagnosis and treatment of different diseases.

The main purpose of this study is to investigate the potential predictive role of the urine proteomics in BP response of patients undergoing RDN. This hypothesis may lead to the emergence of biomarkers in urine of hypertensive patients, in order to optimally select those who will undergo RDN.

This is a prospective observational study enrolling hypertensive patients, aged 18-80 years who will proceed in RDN as participants of randomized control trials. During baseline evaluation HTN diagnosis will be confirmed by office blood pressure measurement (OBPM) and ambulatory blood pressure measurement (ABPM), while urine sample will be collected before RDN for proteomic analysis. The participants will have a follow-up visit in 3 months since baseline procedure for office blood pressure (OBP) and ambulatory blood pressure (ABP) measurements. A cut off value of 5mmHg reduction in ABP or/and 10mmHg reduction in office blood pressure (OBP) on 3 months visit will be set to categorize the patients to responders or non-responders after RDN. The qualitative and quantitative differences of proteins between the two groups of patients will be investigated, based on proteomic analysis results, in order to determine specific urine proteins with predictive role in blood pressure response.

The study results are expected to determine the predictive role of urine proteomics in optimal selection of hypertensive patients who will undergo renal denervation.

DETAILED DESCRIPTION:
Hypertension (HTN) is the most prevalent modifiable risk factor associated with cardiovascular morbidity and mortality, while its prevalence is rising globally. Despite the availability of safe and effective antihypertensive medication, in a large proportion of patients, blood pressure (BP) control to guideline-recommended targets is not achieved. The current knowledge is that sympathetic nervous system hyperactivity contributes to initiation, maintenance and progression of HTN.

Renal denervation (RDN) is a minimally invasive catheter-based method dedicated to disrupt renal sympathetic enervation using different ablation techniques, while is the most extensively investigated device-based therapy for ΗΤΝ. Current endovascular catheter systems access renal arteries and deliver radiofrequency energy, ultrasound energy or use neurotoxic agents such as alcohol, resulting in destruction of the peri-arterial afferent and efferent renal nerves. RDN has experienced ups and downs as a potential treatment option for HTN over recent years of investigation. The initial proof-of-concept, open label clinical trials produced promising results about RDN effectiveness in BP lowering, although, the first randomized sham-controlled trial failed to confirm the previous encouraging results. However, the latest randomized, sham-controlled trials with improved design and methodology demonstrated significant reductions in office blood pressure (OBP) and ambulatory blood pressure (ABP) in patients undergoing RDN. Despite demonstrated efficacy and safety of RDN procedure, about 30% to 40% of patients do not present with a clinically significant BP reduction, even in latest optimally designed clinical trials. This might be due to the pathophysiological substrate in these patients, while identifying a biomarker of BP response could result in a better selection of patients with better response.

The dynamic role of proteins to support the life is documented since the initial stages of biological research. The proteome can be defined as the overall protein content of a biological system such as cell, tissue, biological fluid, etc. Proteomics is the large-scale study of the proteome, as well as the identification and quantification of these proteins. There are some basic steps of proteomic analysis: sample acquisition, protein extraction, protein separation, protein sequence determination and protein identification with bioinformatic techniques in referential databases. Chromatography based techniques are used for protein extraction and high-resolution two-dimensional electrophoresis techniques for proteins separation, while mass spectrometry (MS)-based analysis is widely applied for the protein sequence determination. Proteomic analysis is used in various research settings in detecting diagnostic biomarkers and highlighting pathogenicity mechanisms, alteration of expression patterns in response to different signals or interpretation of functional protein pathways in different diseases. The ultimate goal of proteomics is to better comprehend the molecular complexity while establishing diagnostic and therapeutic healthcare algorithms for the prevention and treatment of diseases.

Α. Aim of the study:

The main purpose of this study is to investigate the potential predictive role of the urine proteomics in BP response of patients undergoing RDN. This hypothesis may lead to the emergence of biomarkers in urine of hypertensive patients in order to optimally select those who will undergo RDN procedure.

B. Study design:

This is a prospective, non-interventional, observational study enrolling a total of 100 patients, with uncontrolled hypertension, treated or untreated, aged 18-80 years, undergoing RDN in the context of randomised clinical trials. During baseline evaluation HTN diagnosis will be confirmed by OBP and ABP measurements, while all patients have to be untreated or treated with maximum of 3 antihypertensive drugs (at least on 50% of maximum dose). Patients with moderate to severe chronic kidney disease (eGFR <45 ml/min), renal artery abnormalities, type I diabetes mellitus and secondary HTN will be excluded. The enrolled cases will have a follow-up visit 3 months after RDN. Data will be collected using a specific form (CRF). These include demographic and somatometric data, past medical history, OBP measurements, ABP measurements, laboratory tests (estimated renal function, serum potassium, serum sodium and serum glucose levels). All patients have to sign an informed consent to participate in the study. Ethics approval has been obtained from the hospital ethical committee board.

C. Methods:

Screen visit: During baseline visit BP will be evaluated with OBP and ABP measurements. Patients with systolic OBP ≥140 mmHg and systolic ABP ≥130 mmHg will be included in the study. The patient profile will include serum tests (glucose, urea, creatinine, sodium, potassium), as well as renal ultrasound in order to exclude anatomic or structural abnormalities of kidneys. Secondary HTN will be excluded, according to HTN guidelines. Urine samples will be collected from all patients and stored in freezer till sending them to Proteomics Research Unit for analyses.

Renal denervation: RDN procedure will be performed 1 to 2 weeks after screen visit by an experienced interventional cardiologist followed by a 1-day hospital stay.

Follow up visit: A follow up visit will be scheduled 3 months after RDN procedure. New OBP and ABP measurements and serum tests (glucose, urea, creatinine, sodium, potassium) will be collected. Data gathering will be completed by statistical analysis. Patients will be categorized as responders or non-responders according to OBP or/and ABP differences between baseline visit and 3 months follow up visit. A 5mmHg reduction in systolic ABP and a 10mmHg reduction in systolic OBP will be set as cut-off values to categorize the patients. At that time point, results from proteomic analyses of baseline urine samples will contribute to the identification of significant qualitative and quantitative differences in proteins between the two groups of patients (responders and non-responders). Information about specific proteins' identity, structure, functions and metabolic pathways in which they are involved, will be collected through biological databases.

Statistical analysis: Normal distribution of all data will be checked with Kolmogorov-Smirnov test. Continuous variables will be expressed as mean and standard deviation (SD), while categorical variables will be presented as percentages (%). Comparisons between categorical variables will be done with χ2 (Pearson's chi-squared test). Comparisons between continuous variables with normal distribution will be done via Student's t-test for unpaired samples, while comparisons between continuous variables which follow non-normal distributions will be done via Mann-Whitney U test. Correlation analysis will be done via Pearson Phi coefficient or Spearman's rho (ρ) based on the distribution of the data set. Statistically significant will be differences with p-value <0.05. Analysis of all data will be performed by SPSS 26 (SPSS Inc, Chicago, Illinois, USA) software.

D. Estimated research outcome:

The study results are expected to determine the predictive role of urine proteomics in blood pressure response of hypertensive patients undergoing renal denervation.

ELIGIBILITY:
Inclusion Criteria:

* All treated patients have to be on standard antihypertensive regimens for at least 8 weeks
* Age 18-80 years
* Office systolic blood pressure ≥140 mmHg and
* Ambulatory systolic blood pressure ≥130 mmHg

Exclusion Criteria:

* eGFR <45mL/min/1.73m2
* Renal artery abnormalities
* Type I diabetes mellitus
* Secondary hypertension
* Pregnant or breastfeeding women
* Psychiatric or neurological disease which does not allow adequate co-operation
* Active cancer on treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, non-interventional, observational study enrolling a total of 100 patients, with uncontrolled hypertension, aged 18-80 years, submitted to renal denervation. During baseline evaluation hypertension diagnosis will be confirmed by OBP and ABP measurememts, while all patients have to be untreated or treated with maximum of 3 antihypertensive drugs (at least on 50% of maximum dose). Patients with moderate to severe chronic kidney disease (eGFR <45 ml/min), renal artery abnormalities, type I diabetes mellitus and secondary hypertension will be excluded. The enrolled cases will be followed up in 3 months after renal denervation. Data will be collected using a specific form (CRF).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Identified proteins' variation rate | 3 months follow up
  In this research protocol the investigators studying urinary proteome changes with potential capacity to predict BP response to RDN procedure. Among the identified proteins in baseline urine, the investigators aim to determine significant proteins' variations between responders and non-responders of BP. Individual proteins will be quantified (μg/g creatinine) by liquid chromatography-mass spectrometry; ELISA and target mass spectrometry analysis will be performed for confirmation. Patients will be classified in responders or non-responders in terms of BP control.

CONTACTS AND LOCATIONS:
Locations (1):
- First Cardiology Clinic, Hippokration General Hospital, National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be available for research purposes under the GDPR regulations.

REFERENCES:
- [Background] Kitt J, Fox R, Tucker KL, McManus RJ. New Approaches in Hypertension Management: a Review of Current and Developing Technologies and Their Potential Impact on Hypertension Care. Curr Hypertens Rep. 2019 Apr 25;21(6):44. doi: 10.1007/s11906-019-0949-4. PMID 31025117
- [Background] Mills KT, Stefanescu A, He J. The global epidemiology of hypertension. Nat Rev Nephrol. 2020 Apr;16(4):223-237. doi: 10.1038/s41581-019-0244-2. Epub 2020 Feb 5. PMID 32024986
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Ng FL, Saxena M, Mahfoud F, Pathak A, Lobo MD. Device-based Therapy for Hypertension. Curr Hypertens Rep. 2016 Aug;18(8):61. doi: 10.1007/s11906-016-0670-5. PMID 27370788
- [Background] Manolis AJ, Poulimenos LE, Kallistratos MS, Gavras I, Gavras H. Sympathetic overactivity in hypertension and cardiovascular disease. Curr Vasc Pharmacol. 2014 Jan;12(1):4-15. doi: 10.2174/15701611113119990140. PMID 23905597
- [Background] Mancia G, Grassi G. The autonomic nervous system and hypertension. Circ Res. 2014 May 23;114(11):1804-14. doi: 10.1161/CIRCRESAHA.114.302524. PMID 24855203
- [Background] Grassi G, Ram VS. Evidence for a critical role of the sympathetic nervous system in hypertension. J Am Soc Hypertens. 2016 May;10(5):457-66. doi: 10.1016/j.jash.2016.02.015. Epub 2016 Mar 4. PMID 27052349
- [Background] Tsioufis C, Kordalis A, Flessas D, Anastasopoulos I, Tsiachris D, Papademetriou V, Stefanadis C. Pathophysiology of resistant hypertension: the role of sympathetic nervous system. Int J Hypertens. 2011 Jan 20;2011:642416. doi: 10.4061/2011/642416. PMID 21331155
- [Background] Laffin LJ, Bakris GL. Hypertension and new treatment approaches targeting the sympathetic nervous system. Curr Opin Pharmacol. 2015 Apr;21:20-4. doi: 10.1016/j.coph.2014.12.006. Epub 2014 Dec 23. PMID 25541034
- [Background] Lauder L, Azizi M, Kirtane AJ, Bohm M, Mahfoud F. Device-based therapies for arterial hypertension. Nat Rev Cardiol. 2020 Oct;17(10):614-628. doi: 10.1038/s41569-020-0364-1. Epub 2020 Apr 14. PMID 32286512
- [Background] SMITHWICK RH. Hypertensive vascular disease; results of and indications for splanchnicectomy. J Chronic Dis. 1955 May;1(5):477-96. doi: 10.1016/0021-9681(55)90061-8. No abstract available. PMID 14367447
- [Background] Liang B, Zhao YX, Gu N. Renal Denervation for Resistant Hypertension: Where Do We Stand? Curr Hypertens Rep. 2020 Sep 3;22(10):83. doi: 10.1007/s11906-020-01094-6. PMID 32880763
- [Background] Schlaich MP, Sobotka PA, Krum H, Lambert E, Esler MD. Renal sympathetic-nerve ablation for uncontrolled hypertension. N Engl J Med. 2009 Aug 27;361(9):932-4. doi: 10.1056/NEJMc0904179. No abstract available. PMID 19710497
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353
- [Background] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Background] Olsen LK, Kamper AL, Svendsen JH, Feldt-Rasmussen B. Renal denervation. Eur J Intern Med. 2015 Mar;26(2):95-105. doi: 10.1016/j.ejim.2015.01.009. Epub 2015 Feb 10. PMID 25676808
- [Background] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939
- [Background] Bakris GL, Townsend RR, Liu M, Cohen SA, D'Agostino R, Flack JM, Kandzari DE, Katzen BT, Leon MB, Mauri L, Negoita M, O'Neill WW, Oparil S, Rocha-Singh K, Bhatt DL; SYMPLICITY HTN-3 Investigators. Impact of renal denervation on 24-hour ambulatory blood pressure: results from SYMPLICITY HTN-3. J Am Coll Cardiol. 2014 Sep 16;64(11):1071-8. doi: 10.1016/j.jacc.2014.05.012. Epub 2014 May 20. PMID 24858423
- [Background] Briasoulis A, Bakris G. Renal Denervation After SYMPLICITY HTN-3: Where Do We Go? Can J Cardiol. 2015 May;31(5):642-8. doi: 10.1016/j.cjca.2014.12.004. Epub 2014 Dec 11. PMID 25828371
- [Background] Townsend RR, Mahfoud F, Kandzari DE, Kario K, Pocock S, Weber MA, Ewen S, Tsioufis K, Tousoulis D, Sharp ASP, Watkinson AF, Schmieder RE, Schmid A, Choi JW, East C, Walton A, Hopper I, Cohen DL, Wilensky R, Lee DP, Ma A, Devireddy CM, Lea JP, Lurz PC, Fengler K, Davies J, Chapman N, Cohen SA, DeBruin V, Fahy M, Jones DE, Rothman M, Bohm M; SPYRAL HTN-OFF MED trial investigators*. Catheter-based renal denervation in patients with uncontrolled hypertension in the absence of antihypertensive medications (SPYRAL HTN-OFF MED): a randomised, sham-controlled, proof-of-concept trial. Lancet. 2017 Nov 11;390(10108):2160-2170. doi: 10.1016/S0140-6736(17)32281-X. Epub 2017 Aug 28. PMID 28859944
- [Background] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589
- [Background] Azizi M, Schmieder RE, Mahfoud F, Weber MA, Daemen J, Davies J, Basile J, Kirtane AJ, Wang Y, Lobo MD, Saxena M, Feyz L, Rader F, Lurz P, Sayer J, Sapoval M, Levy T, Sanghvi K, Abraham J, Sharp ASP, Fisher NDL, Bloch MJ, Reeve-Stoffer H, Coleman L, Mullin C, Mauri L; RADIANCE-HTN Investigators. Endovascular ultrasound renal denervation to treat hypertension (RADIANCE-HTN SOLO): a multicentre, international, single-blind, randomised, sham-controlled trial. Lancet. 2018 Jun 9;391(10137):2335-2345. doi: 10.1016/S0140-6736(18)31082-1. Epub 2018 May 23. PMID 29803590
- [Background] Fengler K, Rommel KP, Blazek S, Besler C, Hartung P, von Roeder M, Petzold M, Winkler S, Hollriegel R, Desch S, Thiele H, Lurz P. A Three-Arm Randomized Trial of Different Renal Denervation Devices and Techniques in Patients With Resistant Hypertension (RADIOSOUND-HTN). Circulation. 2019 Jan 29;139(5):590-600. doi: 10.1161/CIRCULATIONAHA.118.037654. PMID 30586691
- [Background] Bohm M, Kario K, Kandzari DE, Mahfoud F, Weber MA, Schmieder RE, Tsioufis K, Pocock S, Konstantinidis D, Choi JW, East C, Lee DP, Ma A, Ewen S, Cohen DL, Wilensky R, Devireddy CM, Lea J, Schmid A, Weil J, Agdirlioglu T, Reedus D, Jefferson BK, Reyes D, D'Souza R, Sharp ASP, Sharif F, Fahy M, DeBruin V, Cohen SA, Brar S, Townsend RR; SPYRAL HTN-OFF MED Pivotal Investigators. Efficacy of catheter-based renal denervation in the absence of antihypertensive medications (SPYRAL HTN-OFF MED Pivotal): a multicentre, randomised, sham-controlled trial. Lancet. 2020 May 2;395(10234):1444-1451. doi: 10.1016/S0140-6736(20)30554-7. Epub 2020 Mar 29. PMID 32234534
- [Background] Sardar P, Bhatt DL, Kirtane AJ, Kennedy KF, Chatterjee S, Giri J, Soukas PA, White WB, Parikh SA, Aronow HD. Sham-Controlled Randomized Trials of Catheter-Based Renal Denervation in Patients With Hypertension. J Am Coll Cardiol. 2019 Apr 9;73(13):1633-1642. doi: 10.1016/j.jacc.2018.12.082. PMID 30947915
- [Background] Mahfoud F, Azizi M, Ewen S, Pathak A, Ukena C, Blankestijn PJ, Bohm M, Burnier M, Chatellier G, Durand Zaleski I, Grassi G, Joner M, Kandzari DE, Kirtane A, Kjeldsen SE, Lobo MD, Luscher TF, McEvoy JW, Parati G, Rossignol P, Ruilope L, Schlaich MP, Shahzad A, Sharif F, Sharp ASP, Sievert H, Volpe M, Weber MA, Schmieder RE, Tsioufis C, Wijns W. Proceedings from the 3rd European Clinical Consensus Conference for clinical trials in device-based hypertension therapies. Eur Heart J. 2020 Apr 21;41(16):1588-1599. doi: 10.1093/eurheartj/ehaa121. No abstract available. PMID 32211888
- [Background] Arnett DK, Claas SA. Omics of Blood Pressure and Hypertension. Circ Res. 2018 May 11;122(10):1409-1419. doi: 10.1161/CIRCRESAHA.118.311342. PMID 29748366
- [Background] Lam MP, Ping P, Murphy E. Proteomics Research in Cardiovascular Medicine and Biomarker Discovery. J Am Coll Cardiol. 2016 Dec 27;68(25):2819-2830. doi: 10.1016/j.jacc.2016.10.031. PMID 28007144
- [Background] Aslam B, Basit M, Nisar MA, Khurshid M, Rasool MH. Proteomics: Technologies and Their Applications. J Chromatogr Sci. 2017 Feb;55(2):182-196. doi: 10.1093/chromsci/bmw167. Epub 2016 Oct 18. PMID 28087761
- [Background] Zhao M, Li M, Yang Y, Guo Z, Sun Y, Shao C, Li M, Sun W, Gao Y. A comprehensive analysis and annotation of human normal urinary proteome. Sci Rep. 2017 Jun 8;7(1):3024. doi: 10.1038/s41598-017-03226-6. PMID 28596590
- [Background] Loscalzo J. Proteomics in cardiovascular biology and medicine. Circulation. 2003 Jul 29;108(4):380-3. doi: 10.1161/01.CIR.0000079867.56212.17. No abstract available. PMID 12885729
- [Background] Carty DM, Schiffer E, Delles C. Proteomics in hypertension. J Hum Hypertens. 2013 Apr;27(4):211-6. doi: 10.1038/jhh.2012.30. Epub 2012 Aug 9. PMID 22874797
- [Background] Lindsey ML, Mayr M, Gomes AV, Delles C, Arrell DK, Murphy AM, Lange RA, Costello CE, Jin YF, Laskowitz DT, Sam F, Terzic A, Van Eyk J, Srinivas PR; American Heart Association Council on Functional Genomics and Translational Biology, Council on Cardiovascular Disease in the Young, Council on Clinical Cardiology, Council on Cardiovascular and Stroke Nursing, Council on Hypertension, and Stroke Council. Transformative Impact of Proteomics on Cardiovascular Health and Disease: A Scientific Statement From the American Heart Association. Circulation. 2015 Sep 1;132(9):852-72. doi: 10.1161/CIR.0000000000000226. Epub 2015 Jul 20. PMID 26195497